CLINICAL TRIAL: NCT01051817
Title: A Randomized, Multi-center, Double-blind, Proof-of-concept Study to Assess the Effect of Multiple Infusion of AIN457 (10 mg/kg) Versus Placebo on Disease Activity as Measured by MRI Scans Over a 24 Week Period in Patients With Relapsing-remitting Multiple Sclerosis
Brief Title: POC-MD MRI-based Trial in Relapsing-remitting Multiple Scler
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457B2201; 2009-011626-34
Record Dates: First submitted 2010-01-19; First posted 2010-01-20 (Estimated); Results first posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Relapsing-remitting Multiple Sclerosis; RRMS
Keywords: relapsing-remitting multiple sclerosis; RRMS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AIN457 (Experimental)
  Interventions: Drug: AIN457
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AIN457 — infusion 10 mg/Kg
  Arms: AIN457
Drug: Placebo — infusion
  Arms: Placebo

SUMMARY:
A randomized, multi-center, double-blind, proof-of-concept study to assess the effect of multiple infusions of AIN457 (10 mg/kg) versus placebo on disease activity as measured by MRI scans over a 24 week period in patients with relapsing-remitting multiple sclerosis

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2009-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- Czechia (5):
  - Novartis Investigative Site, Hradec Králové, Czech Republic
  - Novartis Investigative Site, Ostrava
  - Novartis Investigative Site, Ostrava-Moravska Ostrava
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Teplice
- Russia (4):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Smolensk
- Ukraine (4):
  - Novartis Investigative Site, Kharkiv
  - Novartis Investigative Site, Kiev
  - Novartis Investigative Site, Odesa
  - Novartis Investigative Site, Vinnitsya

RESULTS

PARTICIPANT FLOW:
Groups:
- AIN457: IV dose 10 mg/kg week 0, 2, 4, 8, 12, 16, and 20.
- Placebo: Placebo IV week 0, 2, 4, 8, 12, 16, and 20.
Period: Overall Study
Arm/Group | AIN457 | Placebo
Started | 38 | 35
Completed | 35 | 26
Not Completed | 3 | 9
Not completed — Adverse Event | 0 | 2
Not completed — Abnormal Test Proceedure reults | 0 | 1
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 | Placebo | Total
Number analyzed (Participants) | 38 | 35 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (9.8) | 32.7 (9.9) | 34.5 (9.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 29 | 50
  Male | 17 | 6 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 35 | 34 | 69
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 36 | 33 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Summary of Raw Number of Cumulative Combined Unique Active Lesions in Patients With Relapsing Remitting Multiple Sclerosis by Visit and Treatment
Description: Combined unique active lesions (CUAL) observed on brain MRI scans performed every 4th week from week 4 to week 24 in patients with relapsing-remitting multiple sclerosis (RRMS). CUAL is defined as: new gadolinium (Gd)-enhancing lesions on T1-weighted, or new or enlarging lesions on T2-weighted MRI scans, without double counting.
Time Frame: weeks 4,8,12,16,20,24,28
Population: Full Analysis Set
Measure: Mean (Full Range); unit: Combined Unique Active Lesions
Groups:
- AIN457B: 10 mg/Kg IV week 0, 2, 4, 8, 12, 16, and 20
Arm/Group | AIN457B | Placebo
Number analyzed (Participants) | 38 | 35
Combined Unique Active Lesions
  Week 4 (n=37,34) | 2.4 [0 to 33] | 3.2 [0 to 16]
  Week 8 (n=36, 31) | 3.9 [0 to 47] | 5.4 [0 to 27]
  Week 12 (n=35,31) | 5.4 [0 to 80] | 8.6 [0 to 34]
  Week 16 (n=32,29) | 6.0 [0 to 104] | 11.5 [0 to 50]
  Week 20 (n=34,27) | 7.7 [0 to 118] | 13.0 [0 to 51]
  Week 24 (n=32,24) | 7.7 [0 to 122] | 15.1 [0 to 64]
  Week 28 (n=32,29) | 9.4 [0 to 142] | 19.9 [0 to 110]

2. Secondary Outcome: Raw Number of Cumulative New Gd-T1 Lesions
Description: The summary of raw number of cumulative new Gadolinium-enhanced T1 lesions observed on brain MRI scans performed every 4th week from WK 4 to WK 28. The end-point is week 24.
Time Frame: MRI brain scans performed every 4 weeks at week 4, 8, 12, 16, 20, 24 and 28 (EOS).
Population: Full analysis set
Measure: Mean (Full Range); unit: cumulative new Gd-T1 lesions
Arm/Group | AIN457B | Placebo
Number analyzed (Participants) | 38 | 35
cumulative new Gd-T1 lesions
  Week 4 (n=37,34) | 1.4 [0 to 31] | 1.7 [0 to 12]
  Week 8 (n= 36,31) | 2.6 [0 to 44] | 3.0 [0 to 16]
  Week 12 (n=35,31) | 4.3 [0 to 76] | 5.5 [0 to 26]
  Week 16 (n= 32,29) | 4.0 [0 to 99] | 7.8 [0 to 36]
  Week 20 (n=34,27) | 5.6 [0 to 112] | 9.2 [0 to 40]
  Week 24 (n=32,24) | 5.4 [0 to 116] | 11.1 [0 to 55]
  Week 28 (n=32,29) | 6.5 [0 to 135] | 14.4 [0 to 99]

3. Secondary Outcome: Raw Number of Cumulative New Gd-T2 Lesions
Description: The summary of raw number of cumulative new Gadolinium-enhanced T2 lesions observed on brain MRI scans performed every 4th week from WK 4 to WK 28. The endpoint is week 24.
Time Frame: MRI brain scans performed every 4 weeks at week 4, 8, 12, 16, 20, 24 and 28 (EOS).
Population: full analysis Set
Measure: Mean (Full Range); unit: Cumulative new Gd-T2 lesions
Arm/Group | AIN457B | Placebo
Number analyzed (Participants) | 38 | 35
Cumulative new Gd-T2 lesions
  Week 4 (n= 37,34) | 2.3 [0 to 30] | 3.1 [0 to 16]
  Week 8 (n=36,31) | 3.6 [0 to 43] | 5.4 [0 to 28]
  Week 12 (n=35,31) | 5.0 [0 to 72] | 8.3 [0 to 34]
  Week 16 (n=32,29) | 5.6 [0 to 91] | 11.0 [0 to 50]
  Week 20 (n= 34,27) | 7.2 [0 to 106] | 12.3 [0 to 51]
  Week 24 (n=32,24) | 7.2 [0 to 110] | 14.6 [0 to 64]
  Week 28 (n=32,29) | 8.8 [0 to 126] | 19.1 [0 to 110]

ADVERSE EVENTS:
Groups:
- PLACEBO: PLACEBO
- AIN457 10mg/kg: AIN457 10mg/kg
Arm/Group | PLACEBO | AIN457 10mg/kg
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/38
Other Adverse Events (participants affected / at risk) | 7/35 | 13/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PLACEBO (N=35) | AIN457 10mg/kg (N=38)
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Oral herpes (Infections and infestations) | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 2
Respiratory tract infection viral (Infections and infestations) | 2 | 2
Viral infection (Infections and infestations) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Headache (Nervous system disorders) | 3 | 1
Paraesthesia (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial